CLINICAL TRIAL: NCT03050203
Title: Surgical Field Custom Pack's Efficacy on Soft Tissue Dissecting Time Reduction, on Relative Risks and Materials Wasted, in Patients Undergoing Spine Surgery: Randomized Controlled Trial
Brief Title: Custom Pack in Spine Surgery
Acronym: kit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0033168
Record Dates: First submitted 2017-02-01; First posted 2017-02-10 (Actual); Results first posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2017-02

CONDITIONS: Bone Diseases; Spine Cancer; Spine Osteoarthritis
MeSH Terms: conditions — Bone Diseases; Spinal Cord Neoplasms; Osteoarthritis, Spine | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- custom pack (Experimental)
  Interventions: Other: custom pack
- standard care (Active Comparator)
  Interventions: Other: standard care

INTERVENTIONS:
Other: custom pack — Preparation of the surgical field using a custom pack. The use of a custom pack provides much of the material provided for the preparation of the surgical field with a single opening of the package , reducing the risk of contamination of the material.
  Arms: custom pack
Other: standard care — The scrub nurse prepares the surgical field opening all the sterile packs it deems necessary for the surgery
  Arms: standard care

SUMMARY:
Recent evidence suggests the efficacy of "custom pack" procedure on the operators reduction time and on the contamination risk due to the opening of many sterile packs. Nevertheless ,the studies available are sponsored by the industry and their results are very few. The aim of this study is to evaluate the correlation and reliability of spine surgery "custom pack" efficacy in adult patients obtained in the reduction of surgery time, relative risks, and materials wasted compared with the standard surgical field procedure practice .

ELIGIBILITY:
Inclusion Criteria:

* Degenerative spinal disease from 2 to 4 levels,
* Oncologic spine disease with only decompression and stabilization.

Exclusion Criteria:

* Revision surgeries,
* Minimally invasive interventions,
* Interventions that provide a dual access, and
* Patients who refuse consent to experimentation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2016-06-16 (Actual); Study Completion 2016-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Nicolini, RN, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Custom Pack | Standard Care
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Custom Pack | Standard Care | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (16.7) | 54.8 (12.4) | 53 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 8 | 10 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
degenerative disease [Count of Participants; unit: Participants] | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Soft Tissue Dissecting Time
Description: minutes from the start of the dissection to complete bone cleaning
Time Frame: up to the first day post intervention
Measure: Mean (Standard Deviation); unit: minues
Arm/Group | Custom Pack | Standard Care
Number analyzed (Participants) | 19 | 18
minues | 38.6 (11.1) | 34 (19.5)

2. Secondary Outcome: Surgery Time
Description: from the incision to the patient's sutures (minutes)
Time Frame: up to the first day post intervention
Reporting Status: Not Posted

3. Secondary Outcome: Postoperative Complications
Description: number of early wound infection
Time Frame: up to 2 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Numbers of Materials Wasted
Description: amount of open sterile materials not used
Time Frame: up to the first day post intervention
Reporting Status: Not Posted

5. Secondary Outcome: Blood Loss
Description: Levels of hemoglobin and hematocrit intraoperative (gas analysis before and after surgery) compared to hemoglobin and hematocrit before surgery and number of blood transfusions both intra- and postoperative.
Time Frame: up to 2 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Pain (Score on the "Numeric Rating Scale")
Description: Pain Score on the "Numeric Rating Scale". The scale had values from 0 to 10 where zero represented no pain and 10 the worst possible pain.
Time Frame: up to the first 3 days post intervention
Reporting Status: Not Posted

7. Secondary Outcome: Length of Stay
Description: number of days spent in hospital
Time Frame: up to 2 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Custom Pack | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes